CLINICAL TRIAL: NCT03852368
Title: UC Reliance# 3107: Exercise and the Brain: Measuring Executive Functions During and Following an Acute Bout of Aerobic Exercise
Brief Title: The Effects of Exercise on Executive Functions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017-3836
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: The Effects of Exercise on Executive Functions
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Effects of Light Exercise in Executive Functions (Experimental): The effects of light exercise in executive functions of adolescents
  Interventions: Other: Exercise
- The Effects of Moderate Exercise in Executive Functions (Experimental): The effects of moderate exercise in executive functions of adolescents
  Interventions: Other: Exercise
- The Effects of Heavy Exercise in Executive Functions (Experimental): The effects of heavy exercise in executive functions of adolescents
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The effects of exercise with different intensity on the executive functions of adolescents

SUMMARY:
The purpose of this research is to develop an assessment protocol that can be used to study the effect of different intensities of exercise on executive functions (EF: attention, working memory, inhibition, and cognitive flexibility). It has been shown that exercise has the potential to improve the development of EF in healthy and special needs children. However, many exercise interventions in the literature lack rigorous control of critical components, such as intensity, making it difficult to draw conclusions about what type and how much exercise might be most beneficial for EF. In addition, to date, no studies have been able to demonstrate the engagement of EF during exercise. This study will focus on developing an assay that measures important self-regulation or EF sub-processes (e.g., attention and inhibitory control) as well as examining engagement of these targets during different exercise intensities. Participants will exercise in different intensities on a cycle ergometer and perform cognitive assessments before, during, and after exercise to evaluate EF. This research will allow us to develop an assessment protocol that can be used in future research to understand the underlying mechanisms underpinning the effects of exercise on EF.

DETAILED DESCRIPTION:
Self-regulation, self-control, and executive functioning are umbrella constructs that encompass processes involved in exerting control over cognitive and behavioral processes. Self-regulation was described as an ability reflecting mature cognition: Mature cognition is characterized by abilities that include being able: (a) to hold information in mind, including complicated representational structures, to mentally manipulate that information and to act on the basis of it, (b) to act on the basis of choice rather than impulse, exercising self-control (or self-regulation) by resisting inappropriate behaviors and responding appropriately, and (c) to quickly and flexibly adapt behavior to changing situations. These abilities are referred to respectively as working memory, inhibition, and cognitive flexibility. Together they are key components of both "cognitive control" and "executive functions…" Some researchers have proposed an integrative framework of self-regulation than encompasses executive functions and self-control. Thus, in this proposal, we have adopted such an integrative framework whereby self-regulation encompasses executive functions, self-control, and other sub-processes. As noted in the specific aims, our meta-analysis and narrative review examining the impact of 28 physical activity (PA) and exercise interventions on EF outcomes in healthy children reported that the targets often shown to improve after exercise were attention, working memory, inhibition, and cognitive flexibility, and preliminary research suggests the strongest effects are on attention and inhibition. The goal of this project is to develop an assay to examine engagement of attention and inhibitory control across several rigorously controlled exercise conditions. This proposal is built on an integrative framework whereby self-regulation encompasses executive functions (EF), self-control, and other sub-processes. Although there is a growing awareness of the benefits of exercise on self-regulatory processes in children including EF, there are still many critical gaps in the research. A recent publication which is a meta-analysis and narrative review examining the impact of 28 physical activity and exercise interventions on EF outcomes in healthy children that highlights some of these gaps. Although earlier results showed that interventions had a significant, small to moderate positive effect on EF, the effects varied widely across studies. This research informed this application in several ways. First, no study demonstrated how or why the interventions improved EF outcomes. Additionally, the behavioral assays or measures varied widely targeting numerous components of EF. The EF targets most often shown to improve after exercise were attention, working memory, inhibition, and cognitive flexibility (each improved in at least five of the included studies). These findings are consistent with recent work at the UC Irvine Pediatric Exercise and Genomics Research Center (PERC); in studies with healthy children and children with special needs, improvements were found after exercise in all four components. Few, if any, studies have been able to demonstrate empirically why participants exhibit improvements in EF after exercise, and studies have not yet demonstrated engagement of EF during exercise. Thus, there is a need to understand why exercise seems to improve these targets. However, the tools used in exercise research to date are limited. Many have been adopted from developmental or educational research, rather than developed specifically to test targets in exercise research; our search yielded only one published measure of self-regulation (cognitive, affective, and motor self-regulation) that has been administered during physical activity. This proposal begins to address these gaps in the literature, by focusing on the development of an assay for important EF targets are improved through exercise and by testing engagement of these targets during exercise of varying intensity

ELIGIBILITY:
Inclusion Criteria:

* Absence of health problems that would preclude participation in exercise
* Male or female between the ages of 10-15 years inclusive at the time of consent
* Minimum level of intellectual functioning, as determined by an IQ (based on cognitive testing) score of 80 or above
* Ability to complete EF testing in English

Exclusion Criteria:

* Other limitations which in the opinion of a physician would preclude ability to perform exercise testing
* Use of illegal drugs or abuse of alcohol based on self-report during screening (this will occur during the one-on-one brief psychological evaluation)
* Pregnancy or breastfeeding based on urine sample test

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
The Effects of Light, Moderate and Heavy Exercise on Attention | 4 weeks
  Attention will be tested with the Hearts and Flowers test
The Effects of Light, Moderate and Heavy Exercise on Working Memory | 4 weeks
  Working Memory will be tested with the Hearts and Flowers test
The Effects of Light, Moderate and Heavy Exercise on Inhibition | 4 weeks
  Inhibition will be tested with Stroop Color-Word test
The Effects of Light, Moderate and Heavy Exercise on Cognitive Flexibility | 4 weeks
  Cognitive Flexibility will be tested with Stroop Color-Word test

SECONDARY OUTCOMES:
The Effects of Light, Moderate and Heavy Exercise on temporal dynamics of executive function processes | 4 weeks
  The temporal dynamics of executive function processes will be measured with EEG/Event-Related Potential (ERP) test

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Exercise and Genomics Research Center, University of California, Irvine, Irvine, California, United States